CLINICAL TRIAL: NCT04822259
Title: A Prospective Multi-Centre Study in Patients Undergoing Total Knee Replacement With JOURNEY II BCS and CR Total Knee System
Brief Title: Evaluate the Performance of JOURNEY II CR and JOURNEY II BCS in TKA Populations
Acronym: JIICRBCSTKA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study design is not reasonable and sponsor decided to terminate the study. No patient enrolled by now
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Journey II CR + BCS.2020.12
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Osteoarthritis; Total knee arthroplasty (TKA); Cruciate Retaining (CR); Bi-cruciate Stabilized (BCS)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- JOURNEY II BCS TKA (Experimental): Undergoing Total Knee Replacement(resurfaced patella) with JOURNEY II BCS Total Knee System
  Interventions: Device: JOURNEY II BCS Total Knee System
- JOURNEY II CR TKA (Experimental): Undergoing Total Knee Replacement(resurfaced patella) with JOURNEY II CR Total Knee System
  Interventions: Device: JOURNEY II CR Total Knee System

INTERVENTIONS:
Device: JOURNEY II BCS Total Knee System — Undergoing Total Knee Replacement(resurfaced patella) with JOURNEY II BCS Total Knee System
  Arms: JOURNEY II BCS TKA
Device: JOURNEY II CR Total Knee System — Undergoing Total Knee Replacement(resurfaced patella) with JOURNEY II CR Total Knee System
  Arms: JOURNEY II CR TKA

SUMMARY:
Background:

The JOURNEY II BCS Total Knee System (JOURNEY II Bi-cruciate Stabilized Total Knee System) consists of femoral component made from oxidized zirconium (OXINIUM)

The JOURNEY II CR Total Knee System (JOURNEY II Cruciate Retaining Total Knee System ) consists of femoral component made from oxidized zirconium (OXINIUM)

Purpose:

Post-market evidence generation for JOURNEY II BCS and JOURNEY II CR Total Knee System

Objectives:

1. Evaluate the performance of JOURNEY II TKA in Asia-Pacific (APAC) patient populations
2. Establish the equivalent performance between JOURNEY II BCS and JOURNEY II CR to support adoption of JOURNEY II CR

Research participants / locations:

A total of at least 176 knees' information will be collected in up to 10 sites. There will be at least eighty-eight (88) knees for JOURNEY II CR TKA group and at least 88 knees for JOURNEY II BCS TKA group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with degenerative osteoarthritis.
* Subject is planning to have bilateral Total Knee Arthroplasty (TKA) using JOURNEY II BCS & CR or have unilateral TKA using JOURNEY II BCS or JOURNEY II CR.*
* Subject is able and willing to provide voluntary consent to study participation.
* Subject is 18-80 years old (inclusive).

[* Bilateral cases can be simultaneous bilateral or staged bilateral (which an interval of 6-8 weeks apart between both knees)]

Exclusion Criteria:

* Subjects with rheumatoid arthritis/inflammatory arthritis, posttraumatic arthritis.
* Previous surgeries including High Tibial Osteotomy (HTO), Unicondylar Knee Arthroplasty (UKA) or Total Knee Arthroplasty (TKA) on the subject knee.
* Subject is pregnant or breast feeding or those at a child-bearing age planning to become pregnant during the follow up.
* Subject does not meet the indication or is contraindicated for JOURNEY II BCS & JOURNEY II CR's Instructions For Use (IFU).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-28 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) at 2 years | 2 years
  The Oxford Knee Score (OKS) is a Patient Reported Outcome (PRO) questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty (TKA). The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.

SECONDARY OUTCOMES:
Forgotten Joint Score (FJS) | 6 months, 1 year , 2 years, 3 years
  The FJS comprises measures for the assessment of joint-specific patient reported outcomes. This questionnaire focuses on the study subject's awareness of the partially or fully replaced knee joint in everyday life. Joint awareness can be simply defined as any unintended perception of a joint. Subjects are asked to rate their awareness of their knee arthroplasty in 12 questions with a five-point Likert response format: "Never", "almost never", "seldom", "sometimes" and "mostly". The item scores are summed and linearly transformed in a 0 to 100 scale with a high value reflecting the ability of the subject to forget about the replaced knee joint during the activities of daily living.
Oxford Knee Score (OKS) | Pre-Operative, 6 months, 1 year, 3 years
  The Oxford Knee Score (OKS) is a Patient Reported Outcome (PRO) questionnaire that was developed to specifically assess the patient's perspective of outcome following Total Knee Arthroplasty (TKA). The OKS is a patient self-completion PRO containing 12 equally weighted questions on activities of daily living. The OKS has been developed and validated specifically to assess perceived function and pain answered on a Likert scale after TKA. Responses to each question ranges from 0-4 with a range of a possible overall score from 0-48. A score of 0 is the worst possible outcome while a score of 48 is the best possible outcome.
Knee Society Score (KSS) | Pre-Operative, 6 months, 1 year, 2 years, 3 years
  The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales:
  1. An "Objective" Knee Score (seven items: 100 points)
  2. A Patient Satisfaction Score (five items: 40 points)
  3. A Patient Expectation Score (three items: 15 points)
  4. A Functional Knee Score (19 items: 100 points)
  The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities. A higher number is a better outcome.
Patient Expectation | Pre-Operative
  The patient expectation will be one single question which have 9 options to choose.
  Patients need to choose at which level of activity he/she expect to recover after surgery.
  The option will be from the most intensive activity to least intensive activity.
Patient Satisfaction | 6 months, 1 year, 2 years, 3 years
  The patient satisfaction will be a corresponding question based on the expectation. It's a five -Likert options (from very satisfied to very dissatisfied) for patients to choose how satisfied he/she is with the surgery to meet the expectation.
Radiographic Assessment | Pre-Operative, 6 months, 1 year, 2 years, 3 years
  Standard radiographic evaluation on antero-posterior (A/P) and lateral views shall be performed at the determined time point before and after surgery in order to identify any radiographic observations such as radiolucent lines around the implant components. The presence of radiolucent lines, osteolysis & implant migration shall be recorded in the electronic Case Report Form (eCRF).
Timed Up and Go Test (TUG) | Pre-Operative, Immediate Post -op to 6 weeks, 6 months, 1 year
  The Timed Up and Go Test assesses mobility, balance, walking ability, and fall risk in adults by measuring time, in seconds, that it takes the individual to stand from a chair, walk a distance of 10 feet (around 3 meters), walk back to the chair, and sit down. The subject will perform the test in their everyday footwear with their walking aid (cane, walker), if applicable [39]. The site will follow the guidelines provided by the Centers for Disease Control and Prevention recording the results on the form provided by the Sponsor
Star Excursion Balance Test (SEBT) | Pre-Operative, Immediate Post -op to 6 weeks, 6 months, 1 year
  The SEBT has been introduced as a simple, reliable, and cost-effective alternative for instrumental devices to assess semi-dynamic balance. The SEBT is a functional test that incorporates a single-leg stance on 1 leg while trying to reach as far as possible with the opposite leg. Each patient performed 3 reaches (trials) in each of the 8 directions. The average of the maximum reach distance in each of the 8 directions was considered for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Yung, Study Director — Smith & Nephew, Inc.
Locations (5):
- China (2):
  - Peking University Third Hospital, Beijing
  - Prince of Wales Hospital, Hong Kong
- India (2):
  - Aster RV Hospital, Bangalore, Bengaluru, Karnataka
  - Noble Hospital & Ruby Hall Clinic, Pune, Maharashtra
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No